CLINICAL TRIAL: NCT03904030
Title: Postoperative Rehabilitation After Knee Arthroplasty, With or Without Anti-Gravity Treadmill
Brief Title: Postoperative Rehabilitation After Knee Arthroplasty: Anti-Gravity Treadmill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orton Orthopaedic Hospital (Other)
Responsible Party: Principal Investigator, Leena Ristolainen, Research Director, Orton Orthopaedic Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OrtonOH
Record Dates: First submitted 2019-04-01; First posted 2019-04-04 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Rehabilitation
Keywords: knee arthroplasty; rehabilitation; anti-gravity treadmill; Randomized study
MeSH Terms: interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: Anti-gravity treadmill rehabilitation and traditional rehabilitation
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-Gravity Treadmill rehabilitation (Experimental): Patients in the intervention group are participating to the Alter G exercises (n=27). The groups are randomized, so after patients have signed consent, an envelop will be opened and there can be seen in which groups patients will participate.
  Interventions: Other: Rehabilitation with or without Anti-Gravity Treadmill
- Traditional rehabilitation (Active Comparator): Traditional exercises with instructions are given to the patients (n=27) (as a control group).
  Interventions: Other: Rehabilitation with or without Anti-Gravity Treadmill

INTERVENTIONS:
Other: Rehabilitation with or without Anti-Gravity Treadmill — The study will include patients with grade III-IV primary knee osteoarthritis. The investigators will take 27 patients to the both groups. The investigators will look after more specifically the anti-gravity treadmill rehabilitation and traditional rehabilitation after arthroplasty. Follow-up is one year. Functional tests will be made and questionnaires will be given to the patients before operation and after operation. After 6 to 8 weeks, 4 months and 12 months of operation questionnaires will be fil up again. After six month the investigators will send a questionnaire and there will be asked possible rehabilitation sessions, use of drugs and possible complications after knee arthroplasty.

SUMMARY:
The aim of this study is to clarify the effectiveness and the usefulness of the anti-gravity treadmill in postoperative rehabilitation after knee arthroplasty. The investigators will compare anti-gravity treadmill rehabilitation and the traditional postoperative rehabilitation with instructions.

The investigators will assume that anti-gravity treadmill exercise after hospitalization will lead to the faster rehabilitation, better walking quality and balance management compared to traditional rehabilitation methods with instructions, where patient themselves do the exercises at home. Additionally, the investigators will assume that quality of life and physical activity will be more increased in the anti-gravity group than in the traditional rehabilitation.

DETAILED DESCRIPTION:
The aim of this study is to clarify the effectiveness and the usefulness of the anti-gravity treadmill in postoperative rehabilitation after knee arthroplasty. This issue is especially relevant because the number of knee arthroplasty patients is increasing. The rehabilitation of knee arthroplasty patients has also appeared to be more challenging than in the case of hip arthroplasty.

The investigators will compare anti-gravity treadmill rehabilitation and the traditional postoperative rehabilitation with instructions. The investigators will recruit the patients either in the anti-gravity group (n=27) or in the traditional rehabilitation (n=27) (randomized study design).

The investigators will assume that anti-gravity treadmill exercise after hospitalization will lead to the faster rehabilitation, better walking quality and balance management compared to the traditional rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* primary knee arthroplasty patients with grade III-V changes

Exclusion Criteria:

* earlier osteotomy to the operated knee
* rheumatoid arthritis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Walking ability | 12 months after operation
  6 minutes walking test will be used
Health-related quality of life | 12 months
  The RAND Health-Related Quality of Life Inventory, RAND 36-Item, will be used, RAND-36 includes: Physical functioning,10 questions; Role functioning/physical, 4 questions; Role functioning/emotional, 3 questions; Energy/fatique, 4 questions, Emotional well-being, 5 questions; Social functioning, 2 questions; Pain, 2 questions; General health, 5 questions; Health change, 1 question. All: 36 questions. Scale: 0 - 100
Perceived pain | 12 months after operation
  Visual analogue scale, (0 to 100, where 0 means no pain at all and 100 means the worst possible pain)

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Hurri, Study Director — Orton Ltd
Locations (1):
- Orton Ltd, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Bugbee WD, Pulido PA, Goldberg T, D'Lima DD. Use of an Anti-Gravity Treadmill for Early Postoperative Rehabilitation After Total Knee Replacement: A Pilot Study to Determine Safety and Feasibility. Am J Orthop (Belle Mead NJ). 2016 May-Jun;45(4):E167-73. PMID 27327921
- [Background] Cheatham SW, Mokha M, Lee M. Postoperative Rehabilitation After Hip Resurfacing: A Systematic Review. J Sport Rehabil. 2016 May;25(2):181-9. doi: 10.1123/jsr.2014-0270. Epub 2015 Jan 22. PMID 25611202
- [Background] Dawson J, Fitzpatrick R, Murray D, Carr A. Questionnaire on the perceptions of patients about total knee replacement. J Bone Joint Surg Br. 1998 Jan;80(1):63-9. doi: 10.1302/0301-620x.80b1.7859. PMID 9460955
- [Background] Freynhagen R, Baron R, Gockel U, Tolle TR. painDETECT: a new screening questionnaire to identify neuropathic components in patients with back pain. Curr Med Res Opin. 2006 Oct;22(10):1911-20. doi: 10.1185/030079906X132488. PMID 17022849
- [Background] Gaudry E, Vagg P, Spielberger CD. Validation of the State-Trait Distinction in Anxiety Research. Multivariate Behav Res. 1975 Jul 1;10(3):331-41. doi: 10.1207/s15327906mbr1003_6. PMID 26829634
- [Background] Guyatt GH, Sullivan MJ, Thompson PJ, Fallen EL, Pugsley SO, Taylor DW, Berman LB. The 6-minute walk: a new measure of exercise capacity in patients with chronic heart failure. Can Med Assoc J. 1985 Apr 15;132(8):919-23. PMID 3978515
- [Background] Konlian C. Aquatic therapy: making a wave in the treatment of low back injuries. Orthop Nurs. 1999 Jan-Feb;18(1):11-8; quiz 19-20. doi: 10.1016/s1361-3111(99)80068-5. PMID 10223000
- [Background] Patil S, Steklov N, Bugbee WD, Goldberg T, Colwell CW Jr, D'Lima DD. Anti-gravity treadmills are effective in reducing knee forces. J Orthop Res. 2013 May;31(5):672-9. doi: 10.1002/jor.22272. Epub 2012 Dec 13. PMID 23239580
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Soininen JV, Paavolainen PO, Gronblad MA, Kaapa EH. Validation study of a Finnish version of the Western Ontario and McMasters University osteoarthritis index. Hip Int. 2008 Apr-Jun;18(2):108-11. doi: 10.1177/112070000801800207. PMID 18645984
- [Background] Valtonen A, Poyhonen T, Sipila S, Heinonen A. Effects of aquatic resistance training on mobility limitation and lower-limb impairments after knee replacement. Arch Phys Med Rehabil. 2010 Jun;91(6):833-9. doi: 10.1016/j.apmr.2010.03.002. PMID 20510971
- [Derived] Jaaskelainen E, Manninen M, Hurri H, Rantasalo M, Zhou Y, Kautiainen H, Ristolainen L. Effectiveness of Anti-Gravity Treadmill Exercise After Total Knee Arthroplasty: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Feb 11;14:e59935. doi: 10.2196/59935. PMID 39932768